CLINICAL TRIAL: NCT04664738
Title: A Phase I Open-Label Trial to Determine the Safety of PEP on a Skin Graft Donor Site Wound
Brief Title: PEP on a Skin Graft Donor Site Wound
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rion Inc. (Industry)
Collaborators: ProPharma Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-00068; 18-004995 (Other: Mayo Clinic)
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-06

CONDITIONS: Skin Graft
Keywords: skin graft; exosome; PEP; wound; healing
MeSH Terms: conditions — Wounds and Injuries | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10 % PEP only (Experimental): Cohort 1: Subjects will receive 10% PEP to the skin graft donor wound.
  Interventions: Biological: 10% PEP
- 20% PEP only (Experimental): Cohort 2: Subjects will receive 20% PEP to the skin graft donor wound
  Interventions: Biological: 20% PEP
- 20% PEP and TISSEEL (Experimental): Cohort 3: Subjects will receive 20% PEP and TISSEEL to the skin graft donor wound.
  Interventions: Drug: TISSEEL; Biological: 20% PEP

INTERVENTIONS:
Biological: 10% PEP — PEP is comprised of platelet derived extracellular vesicles enriched in anti-inflammatory and angiogenic growth factors.
  Arms: 10 % PEP only
Drug: TISSEEL — Fibrin sealant made from pooled human plasma
  Other Names: fibrin sealant
  Arms: 20% PEP and TISSEEL
Biological: 20% PEP — PEP is comprised of platelet derived extracellular vesicles enriched in anti-inflammatory and angiogenic growth factors.
  Arms: 20% PEP and TISSEEL; 20% PEP only

SUMMARY:
The purpose of this study is to determine the safety of a biological therapeutic PEP in participants who have skin graft donor site wounds.

DETAILED DESCRIPTION:
This is an open label phase 1b study of PEP (a leukocyte depleted blood preparation derived from human U.S. sourced pooled apheresed platelets) in patients with at least two donor split-thickness skin graft wounds. One donor site will be treated with the standard post-operative dressing, while the other site will be treated with PEP or PEP+TISSEEL and covered with a standard dressing. TISSEEL is a commercially available fibrin sealant.

ELIGIBILITY:
Main Criteria for Inclusion:

1. Males and females 18-75 years of age.
2. Requiring at least two 20-40 cm2 split-thickness skin grafts by a licensed surgeon or dermatologist
3. Skin graft that meets all the following criteria:

   1. Each graft site has a size of 20-40 cm2 (but can be up to 90 cm2 if found to be clinically indicated during the graft procedure)
   2. Located anywhere on the body (with exception of oral mucosal membranes)
   3. Split-thickness skin graft wound depth of between 8/1000-14/1000 inch
   4. Study donor sites are ≥ 1 cm apart
4. Ability to safely undergo skin graft harvest procedure
5. Capacity to provide informed consent
6. Ability to comply with protocol
7. Subject is judged, by the clinical investigator, to be healthy as evidenced by lack of clinically significant abnormal findings on medical history, physical examination, vital signs, and clinical laboratory tests
8. Subject is able and willing to return to study site for all follow-up visits

Main Criteria for Exclusion:

1. Actively undergoing chemotherapy treatment (localized radiation treatment is allowed if it is not on the skin graft donor site and no active cancer is present)
2. Known history of MRSA (methicillin-resistant Staphylococcus aureus)
3. Known hypersensitivity to aprotinin (Trasylol®)
4. Subjects who are positive for hepatitis B surface antigen (HbsAg), hepatitis C antibody or human immunodeficiency virus (HIV)
5. Any known allergy or sensitivity to adhesive dressings (e.g., Tegaderm)
6. Clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the investigator, not stabilized or may otherwise impact the results of the study
7. Participation in another interventional clinical study or trial in the past 30 days or concurrent participation in another interventional clinical study or trial
8. Subjects with poorly controlled diabetes mellitus (Hemoglobin A1c [HbA1c] ≥ 8%)
9. Subjects with known peripheral neuropathy, or known concomitant vascular problems (such as peripheral artery disease, arterial insufficiency, or venous hypertension) or calciphylaxis
10. Subjects with burns covering ≥ 30% of Total Body Surface Area
11. Currently on or planned to receive hyperbaric wound therapy
12. Pregnant or lactating female subjects
13. Sexually active woman of childbearing potential who is unwilling to use approved contraception method for 3 months after receiving dose of investigational drug
14. Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Acute dose limiting toxicities (DLTs) of PEP / PEP-Tisseel | Up to 2 weeks (within the first 14 days) for each dosing cohort
  The primary endpoint is to determine the acute (within first 14 days) safety and tolerability of PEP or PEP-TISSEEL, as assessed by the occurrence of DLTs on a 20-40 cm2 (but can be up to 90 cm2 if found to be clinically indicated during the graft procedure) skin graft donor site wound at escalating concentrations of PEP delivered at one time point through the 14-day DLT period.
Maximum Tolerated Dose (MTD) of PEP / PEP-Tisseel | Up to 2 weeks (within the first 14 days) for each dosing cohort
  The endpoint is to determine the acute (within first 14 days) safety and tolerability of PEP or PEP-TISSEEL, as assessed by the occurrence of MTDs on a 20-40 cm2 (but can be up to 90 cm2 if found to be clinically indicated during the graft procedure) skin graft donor site wound at escalating concentrations of PEP delivered at one time point through the 14-day MTD period.

SECONDARY OUTCOMES:
Long Term safety of PEP / PEP-Tisseel | 6 months
  The secondary endpoint is to determine the safety and tolerability of a single dose of PEP or PEP-Tisseel delivered at a single time point, as assessed by the occurrence of DLTs through the Day 15-182 DLT period

OTHER OUTCOMES:
Exploratory Endpoint | 6 months
  The exploratory endpoint is to assess wound closure as defined as 100% re-epithelialization after treatment with PEP and PEP-TISSEEL.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sabbah, MD, Study Director — Rion Inc.
Locations (2):
- United States (2):
  - International Research Partners, Doral, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rion company website — https://riontx.com/